CLINICAL TRIAL: NCT01729637
Title: Normothermic Ex-vivo Lung Perfusion: Clinical Experience of the Pressure/Time Curve Profile Study (Stress Index)
Brief Title: SI-EVLP Study: STRESS INDEX in Lung Reconditioning
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD Professor, University of Turin, Italy
Other Study IDs: SI-EVLP
Record Dates: First submitted 2012-11-08; First posted 2012-11-20 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Respiratory Mechanics; Isolated lung perfusion; Ex-vivo lung perfusion; Lung mechanics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to minimize mechanical stress the investigators propose to implement EVLP procedure with a ventilation monitoring guided by the analysis of the Paw-t shape.

DETAILED DESCRIPTION:
Increase of interest about technique of Ex-Vivo Lung Perfusion (EVLP) has highlighted the need of new approaches to respiratory mechanics monitoring to prevent lung stress in atypical physiological settings.

Airway pressure/time curve (Paw-t) shape analysis at constant flow ventilation (Stress Index, SI) is thought to be predictor of lung stress; so the SI coefficient may therefore identify and quantify mechanical stress during ventilation. (1) In experimental studies, the threshold values for SI that best discriminated lungs with signs of Ventilator Induced Lung Injury ranged between 0.9 and 1.1. (2) During EVLP, the isolated lungs are free from the effect of chest wall impairment and represent the effective response of lung parenchyma to ventilatory setting.

Use of SI monitoring in isolated and perfuse lung reconditioning, may be an useful tool to prevent hyperinflation and opening-closing conditions by titrating optimal protective ventilation As previously reported by our group, in the first trial of lung reconditioning, signs of mechanical stress were detected with Paw-t curve. (3) Therefore we implemented EVLP procedure with continuous stress index analysis to detect and quantify the occurrence of hyperinflation or opening closing condition.

ELIGIBILITY:
Inclusion Criteria:

* High risk donor lung, define as:
* the ratio of partial pressure arterial oxygen and fraction of inspired oxygen less than 300
* pulmonary edema
* poor lung deflation or inflation
* blood transfusions exceeding 10 units
* donation after cardiac death as defined by Maastricht category III o IV

Exclusion Criteria:

* donors lung with established pneumonia
* donors lung with severe mechanical lung injury
* donors lung with gross gastric aspiration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: consecutive patient sampling from University Ward of Cardio Surgery of St. Giovanni Battista Hospital of Turin
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Presence of mechanical stress as assessed by analysis of the "Stress Index" | During EVLP procedure (4 hours)
  Stress index is the exponential coefficient of the equation describing the shape of the airway opening pressure vs time (Paw-t) curve during constant flow. This approach is based on the observation that, at constant flow the rate of change of the Paw-t curve corresponds to the rate of change of the compliance of the respiratory system during tidal inflation. A progressive increase in slope (i.e. a downward concavity of the curve) indicates that compliance is progressively increasing with tidal inflation (tidal recruitment). A progressive decrease in slope (i.e. a upward convexity of the curve) indicates that compliance is decreasing with tidal inflation (tidal hyperinflation). Clinical and experimental data show that presence of Stress Index values indicating mechanical stress are associated to morphological, histological and inflammatory evidence of ventilator induce lung injury.

SECONDARY OUTCOMES:
Association between values of Stress Index and occurrence of physiological criteria for EVLP success | During EVLP procedure (4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Paolo Terragni, MD, Principal Investigator — University of Turin - Department of Anesthesia and Intensive Care Medicine
Locations (1):
- University of Turin - Department of Anesthesia and Intensive Care Medicine, Turin, Italy, Italy

REFERENCES:
- [Derived] Terragni PP, Fanelli V, Boffini M, Filippini C, Cappello P, Ricci D, Del Sorbo L, Faggiano C, Brazzi L, Frati G, Venuta F, Mascia L, Rinaldi M, Ranieri VM. Ventilatory Management During Normothermic Ex Vivo Lung Perfusion: Effects on Clinical Outcomes. Transplantation. 2016 May;100(5):1128-35. doi: 10.1097/TP.0000000000000929. PMID 26425874